CLINICAL TRIAL: NCT01568125
Title: Effect of Incretin-related Drugs on Energy and Contents of Dietary Intake in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Incretin-related Drugs on Dietary Intake in Japanese Patients With Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nagaoka Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Kyuzi Kamoi, Investigator, Nagaoka Red Cross Hospital
Other Study IDs: 6
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Incretin-related drugs
  Interventions: Drug: Incretin-related drugs

INTERVENTIONS:
Drug: Incretin-related drugs — DPP-IV inhibitors are administered via per os. GLP-L receptor agonists are administered via subcutaneous injections.
  Other Names: If necessary, other hypoglycemic and insulin drugs

SUMMARY:
It is well known that incretin, particular GLP-１enhances satiety and reduces energy intake in controlling appetite and dietary in humans (Flint A, et al. Gutzwiller JP et al.). Recently, incretin-based therapy has been attracted a lot of interest (Hare KJ, Knop FK). However, it is not clear how the incretin-based therapy affects energy and content of dietary intake in patients with type 2 diabetes mellitus (T2DM). Previously, the investigators reported the amount of energy and content of dietary intake in type 2 diabetic Japanese patients with more than 10 years of long time duration after discovery using questionnaire (Inoue K et al.) and the patients were impaired a secretion of active GLP-1 (Kamoi et al).

The investigators examine whether the incretin-based therapy effects on the energy and content of dietary intake in the same patients before and one year after administration of incretin-related drugs using the same method previously (Inoue K et al.).

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with T2DM without incretin-based therapy, who participated to examine the energy and content of intake using questionnaire reported previously.

Exclusion Criteria:

* Patients with a serious complication in the heart, liver or kidney

  * Pregnant or possibly pregnant patients or lactating patients
  * Patients complicated with a malignant tumor at present.
  * Patients participating in other clinical study.
  * Other than the above, patients judged inappropriate as the subjects of this study by the investigator

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | one year

SECONDARY OUTCOMES:
BMI | One year
Calory of dietary intake | One year
Content of dietary intake | One year

CONTACTS AND LOCATIONS:
Overall Officials: Kyuzi Kamoi, MD, Principal Investigator — Nagaoka Red Cross Hospital; Yoshiko Kontai, RD, Principal Investigator — Universty of Niigata Prefecture; Kanako Inoue, RD, Principal Investigator — Universty of Niigata Prefecture
Locations (1):
- Nagaoka Red Cross Hospital, Nagaoka, Niigata, Japan

REFERENCES:
- [Result] 1. Flint A, et al. Glucagon-like peptide 1 promotes satiety and suppresses energy intake in humans. J Clin Invest. 1998; 101(3):515-520. 2. Gutzwiller JP, et al. Glucagon-like peptide-1: a potent regulator of food intake in humans. Gut. 1999; 44(1):81-86. 3. Verspohl EJ. Novel therapeutics for type 2 diabetes: incretin hormone mimetics (glucagon-like peptide-1 receptor agonists) and dipeptidyl peptidase-4 inhibitors. Pharmacol Ther. 2009; 124(1):113-38. 4. Hare KJ, Knop FK. Incretin-based therapy and type 2 diabetes. Vitam Horm. 2010; 84:389-41 5. Inoue K, Kontai Y, Kamoi K, et al. Energy and content of dietary intake and life related habituation using questionnaire written by Japanese language in Japanese patients with endocrine and metabolism disorders. Abstract in 14 Annual Scientific Meeting of the Metabolism and Clinical Nutrition Society, held at Yokohama of Japan on15th Jan, 2011 (in Japanese).